CLINICAL TRIAL: NCT04648371
Title: Community-based Cognitive Remediation and tDCS to Enhance Seniors' Function and Mental Health
Acronym: CREAtE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: LOFT Community Services (Other)
Responsible Party: Principal Investigator, Angela Golas, Geriatric Psychiatrist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 010/2020
Record Dates: First submitted 2020-11-17; First posted 2020-12-01 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Mental Health Disorder; Aging
Keywords: Cognitive Remediation; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Mental Disorders | interventions — Cognitive Remediation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Centrally administered, computer based generation scheme. Release of assignments only after consent and eligibility, and required baseline data collected. Inability to predict future assignments from past assignments. Creation of an audit trail for the assignment. Balanced Random Assignments to Treatment will be used to generate treatment assignment schedule in a random permuted block design. A file specifying the treatment allocation of each randomization ID will be stored with a member independent of the study. Then, the independent member will access the randomization ID and will access the treatment allocation and program tDCS. The randomization ID will be noted in the CRF but the allocation will not be accessed unless there is an SAE that requires breaking of the blind or the study is complete. In order to ensure that blinding has been maintained, participants and raters will be asked as each patient exits the trial to state what treatment they believe each participant was given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Remediation and Active Transcranial Direct Current Stimulation (Active Comparator): Cognitive Remediation (CR) is a form of group psychosocial intervention that uses a hybrid approach of restorative and strategy based methods to improve areas of cognition (ie. attention, memory, processing speed and learning) through the use of computerized exercises. Transcranial Direct Current Stimulation (tDCS): tDCS will be administered for 30 min/day, at the beginning of each group session. tDCS montage will be frontal with anode placed over Fz and the cathode over Iz. The direct current will be of 2 mA (current density = 0.57 A/m2). CR + tDCS is administered in groups consisting of 2-10 participants and one or two therapists. The groups meet 5 times per week for two hours per session over eight weeks, for a total of 40 sessions in induction phase. Afterwards 3 to 5 sessions per week on monthly boosters.
  Interventions: Other: Cognitive Remediation and Transcranial Direct Current Stimulation
- Cognitive Remediation and Sham Transcranial Direct Current Stimulation (Sham Comparator): CR is identical to the one described under the Active Comparator Arm. However, sham tDCS will consist of active stimulation for only 1 min/day, at the beginning of each group session. tDCS montage and the frequency of the sessions and the boosters will be the same as for the Active Arm.
  Interventions: Other: Cognitive Remediation and Transcranial Direct Current Stimulation

INTERVENTIONS:
Other: Cognitive Remediation and Transcranial Direct Current Stimulation — Cognitive Remediation (CR) is a well-established psychosocial group intervention that aims to improve neurocognitive abilities such as memory performance, executive functioning, processing speed, and attention.
  Transcranial Direct Current Stimulation (tDCS) is a non-invasive brain stimulation method that can be safely administered to awake outpatients. It does not require general anesthesia or surgical implantation. It utilizes low intensity electrical current (e.g., 2 mA) either to increase cortical excitability with an anodal electrode or to suppress cortical excitability with a cathodal electrode.

SUMMARY:
Focusing on seniors with mental health conditions who are living in the community, this initiative proposes to assess the acute and long-term effects of an 8-week course of daily (5 days/week) cognitive remediation (CR) training among 270 participants living in five LOFT senior housing units. The acute course of CR will be followed by monthly one-week boosters until the end of this 5-year study, totaling approximately 24-60 months of follow-up. This trial will also be used as a platform to explore the ability to use transcranial direct current stimulation (tDCS) to optimize response to CR by participant randomization to active versus sham tDCS. Our ultimate goal is to improve the lives of seniors experiencing mental illness and shape a future where they can live independently.

DETAILED DESCRIPTION:
This project requires the complete assessment and treatment of 270 older adult participants living in LOFT senior housing. We will recruit individuals, age 50 or older, who meet criteria for any DSM-V diagnosis, and are living at a LOFT residence.

Prior to enrolment into the study, participants will undergo baseline assessments consisting of clinical, neuropsychological (NP) and functional assessments. Once enrolled, each participant will be randomized to receive transcranial direct current stimulation tDCS (active or sham) concurrent with Cognitive Remediation (CR) for 8 weeks, 5 days per week, followed by 3-5 day of booster sessions on a monthly basis until the end of the study. Trained study staff Personal Support Workers will be administering CR and tDCS for the 8-week intervention phase and the monthly boosters.

Participants will undergo NP and functional assessments at the end of the 8-week induction period, and then on an annual basis until the end of the study.

Primary Aim 1:

To assess whether active-tDCS + CR will result in better cognition (1a), lower fall rates (1b), better function (1c), and less transitions to LTCHs from LOFT (1d) compared to sham-tDCS + CR.

Hypothesis 1a: Participants randomized to active-tDCS + CR will demonstrate better cognition by the end of the 24-60 month follow-up period compared to those randomized to sham-tDCS + CR.

Hypothesis 1b: Participants randomized to active-tDCS + CR will demonstrate lower falls rates by the end of the 24-60 month follow-up period compared to those randomized to sham-tDCS + CR.

Hypothesis 1c: Participants randomized to active-tDCS + CR will demonstrate better self function by the end of the 24-60 month follow-up period compared to those randomized to sham-tDCS + CR.

Hypothesis 1d: Participants randomized to active-tDCS + CR will demonstrate less transitions to Long Term Care Homes by the end of the 24-60 month follow-up period compared to those randomized to sham-tDCS + CR.

Secondary Aim 2:

To build the capacity of LOFT PSWs to deliver tDCS and CR independently and with good fidelity to the intervention model.

Hypothesis 2: At each LOFT location, local PSWs will be certified to deliver tDCS and CR independently by the end of the first year of implementation of the study at each site.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 years and above. The rationale of age cutoff of 50 is that this age is considered a typical geriatric age cutoff especially for people with severe mental illness
2. Any race or ethnicity
3. Any gender identity
4. Meets DSM-V criteria for any disorder
5. Clinically stable as operationalized by (1) having not been admitted to a psychiatric hospital within the 3 months prior to assessment, (2) having had no change in psychotropic medication dosage within the 4 weeks prior to assessment, and (3) ascertained to be clinically and medically stable by one the study psychiatrists.
6. Willingness and ability to speak English
7. Willingness to provide informed consent or assent as applicable.
8. Corrected visual ability that enables reading of newspaper headlines and corrected hearing capacity that is adequate to respond to a raised conversational voice.

Exclusion Criteria:

1. Meets diagnostic criteria for active substance use or dependence within the 6 months prior to the initial assessment except for caffeine or nicotine
2. Electroconvulsive Therapy (ECT) within 6 months of initial assessment
3. Has significant cognitive impairment that, in the opinion of the PI, precludes benefit from CR and therefore study participation.
4. Having any contraindication to tDCS including: the presence of a skin disease, the presence of a pacemaker, implanted brain medical devices, the presence of any metal in the head or suffering from any unstable medical condition or illness that could increase the risk of stimulation (ie. epilepsy)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2026-01-22 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition | Baseline, after 8-week induction phase, and annually until study completion (12, 24, 36, 48, 60 months after baseline)
  Measured by Change in the Montreal Cognitive Assessment (MoCA)(Score range 0-30, higher scores reflect better outcome)
Change in Falls Risk using PPA | Baseline, after 8-week induction phase, and annually until study completion (12, 24, 36, 48, 60 months after baseline)
  Measured by Change in the Physiological Profile Assessment (PPA) (a single index score derived from discriminant function analysis involving weighted scores of independent risk factors relative to a normative database; range: "very low" - "marked" falls risk; high score reflects high falls risk)
Change in Falls Risk using FROP-Com | Baseline, after 8-week induction phase, and annually until study completion (12, 24, 36, 48, 60 months after baseline)
  Measured by Change in the Falls Risk in Older People in the Community (FROP-Com)(Score range 0-60, with higher scores indicative of greater risk)
Change in Functional Performance | Baseline, after 8 week induction phase, and annually until study completion (12, 24, 36, 48, 60 months after baseline)
  Measured by Change in Performance Assessment of Self-Care Skills (PASS). Scale is scored from 0-3, score of 0 indicating inability to complete task, score of 3 indicating ability to complete task independently with no assistance.
Long Term Care Homes Transition | Enrolment to study completion (24, 36, 48, 60 months follow-up period, depending on time of enrolment)
  Measured by Number of Participants who Transition to Long Term Care Homes

SECONDARY OUTCOMES:
Personal Support Workers Delivery of Intervention | Study completion at 60 months
  Number of Personal Support Workers who Completed Training and Able to Administer tDCS + CR Independently

CONTACTS AND LOCATIONS:
Overall Officials: Angela Golas, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: 1. Statistics-Canada. Age and Sex Highlight Tables, 2016 Census. — https://www12.statcan.gc.ca/census-recensement/2016/dp-pd/hlt-fst/as/Table.cfm?Lang=E&T=11.